CLINICAL TRIAL: NCT01675414
Title: Understanding Gastrointestinal Conditions in Children With ASD
Brief Title: Understanding Gastrointestinal Conditions in Children With Autism Spectrum Disorder (ASD)
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Autism Speaks (Other); Columbia University (Other)
Responsible Party: Principal Investigator, Harland S. Winter, MD, Director, Pediatric Inflammatory Bowel Disease Center, Massachusetts General Hospital
Other Study IDs: Grant 2037
Record Dates: First submitted 2012-04-19; First posted 2012-08-30 (Estimated); Last update posted 2012-08-30 (Estimated); Status verified 2012-08

CONDITIONS: Gastrointestinal Disorders; Autism Spectrum Disorders
Keywords: ASD; autism; gastrointestinal; gastrointestinal conditions in children with ASD
MeSH Terms: conditions — Gastrointestinal Diseases; Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: evaluation visit by a pediatric gastroenterologist — medical history, physical exam completed by pediatric gastroenterologist
  Other Names: autism; ASD; pediatric; gastrointestinal

SUMMARY:
The purpose of this research study is to help us learn if children with Autism Spectrum Disorder (ASD) have gastrointestinal (stomach and intestine) problems more frequently than children without ASD do. The investigators hope to learn if children with ASD and gastrointestinal (GI) disorders have certain Problem Behaviors (PB), such as self-injury and aggression, more than children with ASD but no GI disorders do. The investigators want to learn if the Gastrointestinal Symptoms Questionnaire (GIQ) can help us tell which children with ASD also have gastrointestinal disorders.

Hypothesis 1: Children with ASD exhibit high rates of symptomatic GI dysfunction that are not identified by current diagnostic evaluation.

Hypothesis 2: Painful or discomfort-causing gastrointestinal dysfunctions contribute to an elevated incidence or severity of PB in an identifiable subpopulation of PB-expressing children. The investigators anticipate that the proposed study will raise the standard of medical care for children with ASD by improving current methods of identifying GI dysfunction and determining whether there is a significant relationship between GI dysfunction and PB in this population.

ELIGIBILITY:
Inclusion Criteria:

* Children who are ATN Registry subjects between 2 and 17 years old (inclusive)
* Meet criteria for an ASD according to the diagnostic measures Autism Diagnostic Observation Schedule (ADOS) and DSM-IV Symptom Checklist, which were conducted at an established ATN center within the last 18 months

Exclusion Criteria:

* Diagnoses of Rett Syndrome, Childhood Disintegrative Disorder, or other genetic disorders (e.g. Fragile X, Down syndrome, etc.).

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 131 nonselected subjects with ASD
Sampling Method: Probability Sample
Enrollment: 131 (Actual)
Dates: Start 2008-09; Primary Completion 2010-06 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
diagnosis of active gastrointestinal disorder/dysfunction based on the medical history reviewed by and the physical examination performed by a pediatric gastroenterologist | 6 months after initial evaluation by pediatric gastroenterologist

CONTACTS AND LOCATIONS:
Overall Officials: Harland S Winter, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- LADDERS, Massachusetts General Hospital, Boston, Massachusetts, United States